CLINICAL TRIAL: NCT01439308
Title: A Randomized, Double Blind, Placebo Controlled Study to Assessthe Effect of Intranasal Single Dose SB-705498 on the Response Tointranasal Capsaicin Challenge in Non-allergic Rhinitis Patients
Brief Title: Intranasal SB-705498 in Non-allergic Rhinitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111925
Record Dates: First submitted 2011-08-25; First posted 2011-09-23 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis
Keywords: NAR; Capsaicin challenge
MeSH Terms: conditions — Rhinitis | interventions — SB 705498

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Placebo Comparator): 3 incremental capsaicin doses
  Interventions: Drug: Placebo
- Arm 2 (Active Comparator): 3 incremental capsaicin doses
  Interventions: Drug: SB-705498

INTERVENTIONS:
Drug: Placebo — SB-705498 placebo
  Arms: Arm 1
Drug: SB-705498 — 12mg intranasal SB-705498
  Arms: Arm 2

SUMMARY:
This study is designed to look at the affect of SB-705498 on rhinitis symptoms, as induced by capsaicin challenge

ELIGIBILITY:
Inclusion Criteria:

* NAR patients
* Male or female between 18 and 60 years of age inclusive.
* Non-child bearing women or women of child bearing potential if they agree to use contraception as indicated by the protocol
* Non-smoker for at least 6 months with a pack history <5 pack years (Pack years = (No. of cigarettes smoked/day/20) x No. of years smoked).
* Body weight > 50 kg and body mass index (BMI) within the range 19 - 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent.
* Available to complete all the required study measurements.
* Normal 12-lead ECG at screening.
* Subject must demonstrate reactivity to unilateral, intranasal challenge with the selected single dose of capsaicin, defined as development of TSS ≥ 3.
* Normal levels of total plasma IgG and negative allergy skin or Rast test to common aeorallergens.
* Good general health, apart from NAR, as determined by a responsible physician.

Exclusion Criteria:

Past medical history of allergic rhinitis or rhinosinusitis.

* Nasal conditions likely to affect the outcome of the study, i.e. nasal septal perforation, nasal polyps, other nasal malformations.
* A history of gastrointestinal, hepatic, renal or multiple cardiovascular risk factors.
* Positive pre-study drug/alcohol screen.
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for human immunodeficiency virus (HIV) antibody (if determined by the local standard operating procedures (SOPs)).
* History of regular alcohol consumption within 6 months of the study.
* Exposure to more than four new chemical entities within 12 months prior to the start of the study.
* Participation in a clinical trial with a new molecule entity or any other clinical trial within 4 months of the start of the study.
* Use of prescription or non-prescription drugs, as well as of vitamins, herbal and dietary supplements (including St John's Wort) within 2 days prior to each study visit in Part 1 of the study or 14 days prior to the first treatment administration in Part 2 of the study.
* Inability to abstain from all intranasal or oral medication to treat nasal symptoms from the first capsaicin challenge to the completion of the study including: sodium cromoglycate, antihistamines, anticholinergics, alpha-adrenergic agonists and corticosteroids
* History of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* Subjects demonstrating hypersensitivity to the placebo capsaicin challenge at baseline screening.
* Donation of blood or blood products in excess of 500mL within a 56 day period prior the start of Part 2 of this study.
* Pregnant females as determined by positive serum or urine human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Nicotine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* For Part 2 only: Subjects with known lactose intolerance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Assessment of total symptom score (TSS) after unilateral, incremental dose, intranasal challenge with capsaicin | 0-4hours following dosing
Assessment of total Ipsilateral secretion's weight after unilateral, incremental dose, intranasal challenge with capsaicin | 0-4hours following dosing

SECONDARY OUTCOMES:
Change from baseline in peak nasal inspiratory flow (PNIF) after unilateral, incremental dose, intranasal challenge with capsaicin | 0-4hours following dosing
Assessment of Total Contralateral secretion's weight after unilateral, incremental dose, intranasal challenge with capsaicin | 0-4hours following dosing
Number of participants with Individual Symptoms as assessed by TSS components after unilateral, incremental dose, intranasal challenge with capsaicin | 0-4hours
Soluble biochemical mediators, including but not limited to neuropeptides, in nasal secretions induced after unilateral, incremental dose, intranasal challenge with capsaicin | 0-4hours following dosing
Intranasal, single dose SB-705498 plasma PK parameters-Cmax | 0-4hours
Intranasal, single dose SB-705498 plasma PK parameters- Tmax | 0-4hours post dosing
Intranasal, single dose SB-705498 plasma PK parameters- AUC(0-t) | 0-4hours post dosing
Number of participants with adverse events | Day 1
Number of participants with vital signs data outside range of potential clinical importance- Systolic blood pressure (SBP) and diastolic blood pressure (DBP) | Day 1
Heart rate | Day 1
Number of participants with nasal examination data | Day 1
Number of participants with abnormal ECG findings | Day 1
Body temperature | Day 1
Number of participants with abnormal hematology values | Day 1
Number of participants with abnormal clinical chemistry values- Carbon dioxide content/Bicarbonate, Cholesterol, Potassium, Triglycerides | Day 1
Number of participants with abnormal clinical chemistry values- Creatinine | Day 1
Number of participants with abnormal clinical chemistry values- Gamma Glutamyl Transferase, Lactate Dehydrogenase | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 111925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register